CLINICAL TRIAL: NCT05116059
Title: To Evaluate the Efficacy and Safety of Amphotericin B Colloidal Dispersion (ABCD) in the Treatment of Invasive Fungal Disease: a Multicenter, Retrospective, Observational, Non-interventional Registration Study
Brief Title: To Evaluate the Efficacy and Safety of ABCD in the Treatment of IFD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSPC-ABCD-K02
Record Dates: First submitted 2021-10-12; First posted 2021-11-10 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Invasive Fungal Disease
Keywords: Amphotericin B Colloidal Dispersion; Invasive fungal disease
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amphotericin B colloidal dispersion（ABCD） — The dosage and course of ABCD were determined by clinicians, and this study was registered according to clinical practice

SUMMARY:
In order to better guide clinical medication, verify the efficacy and safety of ABCD in the treatment of various invasive fungal disease, the investigators have designed a multi-center, retrospective registration study. Diagnosis and treatment data for patients with different types of invasive fungal disease in clinical actual environment was collapsed by a database for collaborative exchange on antifungal research.

DETAILED DESCRIPTION:
This study is a retrospective, non-interventional, and observational study. The clinical data of the patient during hospitalization shall be collected at least 2 weeks after the end of the ABCD drug, including basic data of the patient, laboratory data and clinical treatment, mainly covering antifungal medications, such as pretreatment measures, drug dosage and dispensing method, route of administration, duration of administration, efficacy and adverse reactions, etc. If adverse events related to ABCD have not ended after 2 weeks, investigators are advised to follow up until the adverse events recover or stabilize. It is hoped that the basic situation of Chinese invasive fungal patients is described, and ABCD is evaluated in the treatment of invasive fungal patients. In addition, prognostic factors can be analyzed to optimize clinical medication regimen and provide basis support for clinical medication of ABCD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients with possible/probable/proven invasive fungal disease according to EORTC-MSG diagnostic criteria.
3. Patients received ABCD alone or in combination with other antifungals on either empirical, diagnosis-driven or targeted therapy.
4. There is no limit to the patient's previous treatment plan.

Exclusion Criteria:

1. Patients judged by clinicians to be unsuitable for this study.
2. Patients with incomplete data or other factors affecting the judgment of efficacy and safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive fungal disease and accepted of ABCD
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
therapeutic response rate | within one week of the last administration of ABCD
  Patients with hematological tumors are evaluated for efficacy according to the diagnostic criteria and treatment principles for invasive mycoses in patients with hematological diseases/malignant tumors (the sixth revised edition). Efficacy assessment criteria for patients with non-hematological tumors are defined as complete and partial response as effective, and stable, progress and death as ineffective.
Infusion reaction, renal toxicity, hypokalemia, liver function and other adverse events [Safety and Tolerability] | from the date of start medication until the date of last dose of ABCD. If the adverse reaction has not ended after 2 weeks, clinicians are advised to follow up until the adverse event has recovered or stabilized (Assessed up to 1 week).
  The incidence, start and end times, and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: zhengyin Liu, PhD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Zhang Q, Ma W, Chu ZB, Xu L, Xing H, Wang J, Lin J, Liu Z. Efficacy and Safety of Amphotericin B Colloidal Dispersion for Patients with Invasive Fungal Disease and Febrile Neutropenia: A Registry-Based, Multicenter, Retrospective, Real-World Study. Infect Drug Resist. 2025 May 13;18:2475-2487. doi: 10.2147/IDR.S494985. eCollection 2025. PMID 40384797